CLINICAL TRIAL: NCT05289700
Title: Multicentric, Double-blind, Randomised Controled Trial of Hyperbaric-oxygen Therapy (HBOT) Versus Placebo for Treating Vaso-Occlusive Crisis (VOC) in Sickle Cell Disease (SCD) After 8 Years Old
Brief Title: Hyperbaric-oxygen Therapy (HBOT) Versus Placebo for Treating Vaso-Occlusive Crisis (VOC) in Sickle Cell Disease (SCD)
Acronym: HBOT-SCD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: University Hospital, Toulouse (Other); Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Jerome Stirnemann, Assistant Head of the Internal medicine Unit, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-01707
Record Dates: First submitted 2022-02-04; First posted 2022-03-21 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Sickle Cell Disease; Hyperbaric Oxygen Therapy; Vaso-occlusive Crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Intervention is a treatment with Hyperbaric Oxygen Therapy in Hyperbaric chamber. Placebo is entry in hyperbaric chamber but without oxygen and with a minimal pression. Within 4 hrs (or at the latest 12 hrs) of their initial consultation at their hospital's ED, patients who have agreed to participate in the study will be randomised between the HBOT intervention group (2 ATA, 95 min, FIO2=1) and the placebo group (1.3 ATA, 95 min, FIO2=0.21). Patients undergo a first session (HBOT/placebo) in the hyperbaric chamber and then return to their ward.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomisation will be double-blinded: neither the patient nor physician caring for the patient will be informed of the strategy. Only the Hyperbaric Chamber team, in charge of the session, will be informed of the treatment arm which has been attributed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBOT intervention group (2 ATA, 95 min, FIO2=1) (Experimental): Hyperbaric Oxygen Therapy (HBOT) is the administration of oxygen at a pressure higher than atmospheric pressure (2 ATA). By breathing pure oxygen at twice the atmospheric pressure, its concentration in the blood is multiplied by nearly ten times. This allows a greater oxygen concentration in poorly vascularised areas of the body.
  Interventions: Device: HBOT in Hyperbaric chamber
- placebo group (1.3 ATA, 95 min, FIO2=0.21) (Placebo Comparator): Hyperbaric chamber is the same chamber used for HBOT, but with a limited hyperpressure (1.3 ATA) and using ambient air (FIO2=0.21), with illusion of treatment in healthy volunteers.
  Interventions: Device: Hyperbaric chamber for placebo

INTERVENTIONS:
Device: HBOT in Hyperbaric chamber — HBOT is the administration of oxygen (FIO2 = 100%) at a pressure higher than atmospheric pressure (2 ATA). The pressure increase is achieved by introducing compressed air into the hyperbaric chamber. This study will use a hyperbaric chamber that is already marketed, licensed and used in other diseases.
  Other Names: Hyperbaric Oxygen Therapy
  Arms: HBOT intervention group (2 ATA, 95 min, FIO2=1)
Device: Hyperbaric chamber for placebo — Hyperbaric chamber is the same chamber used for HBOT, but here with a limited hyperpressure (1.3 ATA) and using ambient air (FIO2=0.21), with illusion of treatment in healthy volunteers. All other aspects of the procedure are identical to those of the intervention. As in the intervention arm, there will be a compression period (although shorter), of 5 min, followed by 85 min at 1.3 ATA, then a decompression period of 5 min (total duration of 95 min).
  Other Names: Placebo Comparator
  Arms: placebo group (1.3 ATA, 95 min, FIO2=0.21)

SUMMARY:
This is a randomised, controlled, double-blind, placebo trial of HBOT (intervention) superiority in the treatment of VOC in SCD, to demonstrate the effectiveness of HBOT for the decrease in pain level in the treatment of SCD-VOC.

DETAILED DESCRIPTION:
Background: Sickle cell disease (SCD) is one of the most common genetic diseases in the world, affecting approximately 310,000 births each year and causing >100,000 deaths. Vaso-occlusive crisis (VOC) is the most frequent complication of SCD, leading to bone pain, thoracic pain and/or abdominal spasms and is the main cause of death in patients with SCD. It is linked to sickling which is often triggered by internal and external environmental conditions such as acidosis, cold, dehydration, hyperthermia, infection and especially hypoxia. Sickling is initially reversible if local oxygenation supply and conditions are improved.

Rationale: The use of hyperbaric oxygen therapy (HBOT) should enable the patient's tissues to receive the extra oxygen necessary by increasing the amount of dissolved O2 in blood which in turn would limit sickling. A pilot study of 9 patients showed the potential positive effects of HBOT on VOC induced pain. International guidelines indicate that SCD-induced VOC is one of the potential indications for HBOT, even though the evidence available is weak.

Aim and objectives: To demonstrate the analgesic effect of HBOT for VOC and to analyse the procedure's safety, impact on the biological markers of SCD-induced VOC, progression of SCD and cost-effectiveness.

Methodology: This study will be a multicentric, double-blind, randomised controlled trial. Any patient presenting at one of the participating centres' Emergency Departments (EDs) with VOC is eligible to be evaluated, included and randomized. Inclusion criteria: Patients aged 8 years or over with a major SCD, having a VOC non-responsive to level 2 analgesics (WHO classification), with or without Acute Chest Syndrome (ACS). Exclusion criteria: Pregnancy, indication for artificial ventilation, proven contraindication for HBO, blood velocity > 200 cm/sec previously measured with transcranial Doppler, previous history of stroke, patient requiring more than 2 l/min of normobaric oxygen in order to achieve an SpO2 (peripheral oxygen saturation) ≥ 92%. Patients with exclusion criteria, although precluded from the randomisation process, will however be eligible to undergo the HBOT intervention and become part of the cohort. Measurements and procedures: In all cases, included patients will receive usual care for VOC, including hydration, analgesics (patient-controlled analgesia with morphine), normobaric oxygen therapy and where medically indicated, antibiotic therapy and/or transfusions. Within 4 to 12 hours of their initial consultation at their hospital's ED, patients who have agreed to participate in the study will be randomised between the HBOT intervention group (2 Atmosphere Absolute pressure [ATA], 95 min, FIO2 = 1) and the placebo group (1.3 ATA, 95 min, FIO2 = 0.21). Patients will undergo a first session in the hyperbaric chamber and then return to their ward. The second (and third) session (for both groups) will systematically take place within 24 h (max. 36 h) of the first session. If the visual analogue scale (VAS) pain score is ≤ 2 without the use of level 3 analgesics at the standard dosage, subsequent sessions will be cancelled. Difference in the visual analogue scale (VAS) pain score before and after HBOT and other outcomes will be compared between the intervention and placebo groups. A superiority of HBOT compared placebo group in VOC should be demonstrated, with decrease of pain, length of stay and cost.

Expected results and their impact: Expected benefits of HBOT are the reduction of: pain experienced, duration of the crisis, number of transfusions required, the number of morphine doses, reduction of length of stay and reduction in the frequency of ACSs and VOCs.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8 or over;
* Diagnosed with a major SCD disorder (SS, SC, Hb O Arab, Sβ0 and Sβ+ -thalassemias);
* Presentation of a Vaso-Occlusive Crisis (VOC), with or without Acute Chest Syndrome,
* Unresponsive to level 2 analgesics (WHO classification)
* Which fulfils the criteria necessary for consultation at an ED;
* Ability to carry out the Valsalva manoeuvre;
* Ability to give informed consent and sign a written informed consent form (consent and signature of legal guardian authorised).

Exclusion Criteria:

* Pregnancy;
* Indication for artificial ventilation (non-invasive ventilation/oro-tracheal intubation);
* Proven contraindication for HBOT established by a physician responsible for hyperbaric medicine;
* Anomaly in the results of prior transcranial Doppler (TCD) ultrasound (> 200 cm/sec) or a previous history of stroke (but TCD will not be performed for the study);
* Patients requiring more than 2 l/min of normobaric oxygen in order to maintain an SpO2 ≥ 92%.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of visual analogue scale (VAS) pain score | Baseline (before HBOT session ; H0) and 6th hour after the start of the HBOT session (H6)
  The visual analog scale (VAS) pain score is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain" (10). Change = (Hour 6 VAS score - Baseline VAS score) ; Difference in the global visual analogue scale (VAS) pain score evaluated immediately before (in the ED ; H0) and 6 hrs after (on the ward) the HBO therapy/placebo session (H6).
Change from baseline of a number of patients with composite outcome (VAS pain score >4 and/or mean morphine dosage > 1mg/h IV) | Baseline (before HBOT session ; H0) and 6th hour after the start of the HBOT session (H6)
  The visual analog scale (VAS) pain score is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain" (10). Change = Number of patient with composite score at H6 - Number of patient with composite score at H0.

SECONDARY OUTCOMES:
Change from baseline of the mean morphine dosage treatment (mg/h IV) at H6 | Baseline (before HBOT session ; H0) and 6th hour after the start of the HBOT session (H6)
  Change in mean hourly concentration dosage of morphine between the mean concentration before HBOT Session (H0) and the mean concentration during the 4 hours after session (H6) [morphine concentration during session (2 hours) is not included in the calculation]. In case of treatment with oral morphine, an equivalent of IV doses will be used.
Change from baseline of the mean morphine dosage treatment (mg/h IV) at H24 | Baseline (before HBOT session ; H0) and 24th hour after the start of the HBOT session (H24)
  Change in mean hourly concentration dosage of morphine between the mean concentration before HBOT Session (H0) and the mean concentration during the 22 hours after session (H24) [morphine concentration during session (2 hours) is not included in the calculation]. In case of treatment with oral morphine, an equivalent of IV doses will be used.
time to discontinuation of IV opioids | From admission date until discharge date (up to 1 month)
  Time between admission and discontinuation of intra-venous opioids, during hospitalisation before discharge and/or rehabilitation transfer
length of hospital stay | From admission date until discharge date (up to 1 month)
  Number of days between admission and hospital discharge
Number of patients experiencing relief from pain (ie reduction of VAS>30%) at Hour 6 | 6th hour after the start of the HBOT session (H6)
  The visual analog scale (VAS) pain score is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain" (10). Number of patient with decreasing of VAS pain score>30% between Hour 6 and baseline (before HBOT session ; H0).
Number of patients experiencing relief from pain (ie reduction of VAS>30%) at Hour 24 | 24th hour after the start of the HBOT session (H24)
  The visual analog scale (VAS) pain score is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain" (10). Number of patient with decreasing of VAS pain score>30% between Hour 24 and baseline (before HBOT session ; H0)

OTHER OUTCOMES:
Patient's "global impression of change" | 6th hour (H6) and 24th hour (H24) after the start of the HBOT session
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
time until end of VOC (Vaso-occlusive crisis) | From admission date until discharge date (up to 1 month)
  Time (number of hours) until VOC is finished. VOC is terminated when VAS<2, in the absence of painkillers of level III. The visual analog scale (VAS) pain score is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain" (10).
Number of transfusion therapies during hospitalization | From admission date until discharge date (up to 1 month)
  indications for and implementation of transfusion therapies during hospitalization
Number and type of complications | From inclusion date, up to one year after baseline (HBOT session)
  notably Acute Chest Syndrome, priapism, stroke or other
Lactate Dehydrogenase dosage in blood sample | From admission date until discharge date (up to 1 month)
  In unit/L. reported at each dosage, during hospitalisation
C-reactive protein (CRP) in blood sample | From admission date until discharge date (up to 1 month)
  In mg/L
Number of patients with readiness discharge | From admission date until discharge date (up to 1 month)
  readiness for discharge as judged by the patient or physician
Number of new hospitalisations | During one year after hospitalisation
  further hospitalisations during the following year
treatment costs | From admission date until discharge date (up to 1 month)
  Cost of the strategy with HBOT session or placebo
Number of patients with death | During one year after hospitalisation
  death during hospitalization or after discharge

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - Hospices civils de Lyon, Lyon
  - Centre de compétences Sd drépanocytaires, Toulouse
- HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No